CLINICAL TRIAL: NCT04311203
Title: Evaluation of Mental Health First Aid From the Perspective of Workplace End Users - EMPOWER: Protocol of Trial Phase
Brief Title: Evaluation of Mental Health First Aid From the Perspective of Workplace End Users
Acronym: EMPOWER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London South Bank University (Other)
Collaborators: Mental Health First Aid England (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Evaluation of MHFA
Record Dates: First submitted 2020-03-03; First posted 2020-03-17 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Help-Seeking Behavior
Keywords: Mental health first aid; Help-seeking behaviours; Workplace; Process evaluation; Economic evaluation
MeSH Terms: conditions — Help-Seeking Behavior

STUDY DESIGN:
Intervention Model Description: The study is a multi-centred, two-arm clustered randomised controlled trial. Organisations will be randomly allocated to the control or intervention. The intervention is the standard MHFA intervention provided by Mental Health First Aid England (MHFAE). The control condition will be organisations having a brief consultation from MHFAE on promoting mental health and well-being in the workplace.
Masking Description: Participants and researchers will not be blinded to treatment allocation due to the nature of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health First Aid Intervention (Experimental): Two-day MHFA training provided by MHFA England. Organisations will raise awareness of the presence of MHFA in the workplace, with delivery of MHFA by trained members to participants in the workplace.
  Interventions: Behavioral: Mental Health First Aid
- Control (No Intervention): A brief consultation from MHFAE on the promotion of mental health and well-being in the workplace.

INTERVENTIONS:
Behavioral: Mental Health First Aid — The intervention has 3 parts:1.Two-day MHFA training provided by MHFA England. A manualised programme designed to provide individuals with: an in-depth understanding of mental health and the factors that can affect wellbeing, practical skills to spot triggers and signs of mental health issues, confidence to step in, reassure and support a person in distress, enhanced interpersonal skills such as non-judgemental listening, knowledge to help someone recover their health by guiding them to further support - whether that's self-help resources, through their employer, the NHS, or a mix. 2.Raising awareness of the presence of MHFA in the organisation. 3.The application of MHFA to participants in the workplace using the manualised five-stage approach, ALGEE: Approach the person, assess and assist with any crisis; Listen and communicate non-judgementally; Give support and information; Encourage the person to get appropriate professional help and Encourage them to seek other forms of support.
  Arms: Mental Health First Aid Intervention

SUMMARY:
This trial will evaluate the effectiveness of Mental Health First Aid in the workplace. Half of the organisations will receive Mental Health First Aid training and half will receive treatment as usual (a brief consultation from Mental health First Aid England on mental health and well-being in the workplace).

DETAILED DESCRIPTION:
The EMPOWER study will implement a cluster randomised controlled trial (cRCT) to examine the effectiveness and cost-effectiveness of MHFA in the workplace on help-seeking behaviours of employees, with embedded qualitative, process and social impact evaluations . In order to best answer questions regarding effectiveness, mechanisms and acceptability/feasibility, a design combining a RCT with a qualitative component will be adopted. The qualitative component will assess the efficiency, utility, usability, feasibility, acceptability as well as the mechanisms underlying the intervention. This registration details the trial element of EMPOWER only.

Data will be collected from employees working in eligible UK organisations expressing an interest to MHFAE in undertaking MHFA training. Organisations expressing an interest (directly to MHFAE), who are willing to take part in the study will be asked to contact Graham Durcan (Centre for Mental Health) for detailed information about the study. If willing to take part, organisations will sign a written agreement and their contact details will be sent to the research team. The research team will email the lead contact, detailing what will happen next, asking for company demographics and requesting organisations send a standard email to ALL employees providing information about the study with a link to the survey for completion of baseline measures. Consent will be sought, using Qualtrics, before completing the online survey. One, two and three weeks later the research team will send the organisation lead another standard email, to be sent to all employees, as a gentle reminder to complete the survey. After this period, participants who have not completed the survey will be treated as lost to follow-up.

Organisations will be assigned randomly to the intervention or control arm after completing baseline measures, using computer-generated random numbers through Random.org:

https://www.random.org/randomness/. An independent researcher not associated with the study will generate the random sequence and communicate this via email to the research team. The unit of randomisation is organisation and randomisation of organisations will be stratified by size of organisation, with three strata being defined22, small (< 50 employees), medium (50-249 employees) and large (> 250 employees).

To optimize completion of follow-up measures, at each follow-up point the research team will send organisations up to four weekly email reminders to ask employees to complete measures.

Participant data will be exported from Qualtrics into SPSS version 22 by the research team (and any hard copies entered manually), stored on a password-protected network drive, will be accessible only to research team members and will only be linked directly with their participant ID code. Any hard copies of data will be destroyed by confidential waste disposal fifteen years after the research findings have been published. Electronic copies of data will be stored in two archives. In both cases, only anonymous data will be archived at London South Bank University archive and a national data repository.

Data monitoring will be conducted by the Trial Steering Committee (TSC) comprising a trialist, statistician and health economist and will act as Data Safety Monitoring Board (DSMB). The TSC will oversee the conduct of the trial independently of and on behalf of the project funders and sponsors and ensure it is carried out with reference to good practice. The TSC will have ultimate responsibility for deciding if the trial should be stopped on grounds of efficacy. The TSC is a sub-group of the project Expert Reference Group (ERG) set up by the funders, and will audit the trial conduct through reports submitted to it by the researchers on a three-monthly basis'

We anticipate little risk to participants in the study. The Senior Manager in each company will be asked to report to the CI in writing any adverse or untoward incidents that occur because of the study. The CI will assess each adverse event and decide on an appropriate course of action. In case of Serious Adverse Events (SAEs), i.e. those causing serious injury or death, the CI will notify the Ethics Committee and the TSC as soon as possible after being notified. A TSC within the ERG consisting of members independent of the investigators, their employing organisations, funders and sponsor will monitor trial progress and conduct and will have ultimate responsibility for deciding if the trial should be stopped on the grounds of safety.

The sample size calculation is based on a simplification of the proposed analysis model.

To be able to detect a change of two additional help seeking resources11, with 80% power at the 0.05 alpha level, assuming that the mean in the control group is 1 and in the intervention group 3 with a common standard deviation of 8, 506 participants are required, increasing to 596 allowing for 15% attrition at 6 months. Pilot data indicates a response rate of 40% across organisations and an average cluster size of 72 employees (calculated from organisations currently signed up) therefore approximately 29 employees per organisation (cluster size). With 24 clusters, 12 organisations per condition, and assuming an intraclass correlation coefficient (ICC) equal to 0.01 (ICC's are lower for participant outcomes as opposed to process variables, when cluster size is large and when estimates are adjusted by participant baseline characteristics21) a minimum target sample size is 763, rounded up to 800, 400 per condition

All outcomes will be described with the appropriate descriptive statistics: mean and standard deviation for continuous outcomes (or medians and interquartile range for skewed data), and counts and percentages for dichotomous and categorical outcomes.

The analysis of the primary outcome will estimate the mean difference (with 95% confidence intervals) in the Actual Help-Seeking score at 6-month follow-up between the intervention (MHFA) and standard care groups using a mixed effects repeated measures model (which assumes incomplete outcome data to be missing at random). The model will incorporate demographic and other baseline covariates as fixed effects. The dependent variable will be the count of help sources on the Actual Help-Seeking questionnaire. The independent variable will be 'time point'. The effect size of the intervention will be estimated as the exponentiated coefficient for the interaction term between time-point (baseline versus 6-months follow-up) and intervention status (MHFA versus control group). A random effect of participant will be included in the model to adjust for the repeated measures on participants. 'Employing organisation' will be included as a higher level random effect (with participants nested in employers). Statistical significance will be at the 5% level.

Secondary outcomes will be analysed using an appropriate generalised linear model, for example binary logistic regression for dichotomous outcomes and ordinal logistic regression for ordered categorical outcomes. All models will be adjusted for employing organisation and baseline score (where applicable).

Age, gender, level of education, ethnicity, nature and frequency of and MHFA interventions directly experienced will be included in the primary analysis as covariates.

The missing at random assumption for primary outcome data will be assessed further in sensitivity analyses. Treatment effects will be estimated under varying assumptions of data being missing not at random using pattern-mixture models. A complete case analysis will also be conducted.

Graham Durcan from The Centre for Mental Health (CMH) has oversight of the project management on behalf of the funders. The Chief Investigator [CI] (Callaghan) has overall responsibility for the research.

A Research Management Group (RMG), which the CI will chair, comprising all authors, will advise and assist on the project's management. The RMG meets every 6 weeks.

An Expert Reference Group (ERG), a group of independent research experts and lay people and the CI, will provide subject matter expertise to the funders and work with the CMH and London South Bank University's representatives to guide and oversee the impact of the research. The ERG meets quarterly for the entirety of the project's duration.

ELIGIBILITY:
Inclusion Criteria: organisations expressing an interest (directly to MHFAE) in undertaking MHFA training, who have not undertaken this training previously; organisations who agree to participate and are able to provide data on sickness absenteeism, presenteeism and other productivity data

Exclusion Criteria: organisations who have already introduced MHFA across all sites and departments; those who decline to participate in adopting MHFA training; organisations and employees who participated in the pilot study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in Employees' help-seeking behaviour | 6, 12 and 24 months.
  Measured by the Actual Help-Seeking Questionnaire [AHSQ] (Rickwood et al., 2005).The AHSQ measures help-seeking behaviour in the two-weeks preceding the assessment. Help-seeking behaviour is determined by listing the number of help sources and whether these have been sought in the time period and the issue for which they have been approached.

SECONDARY OUTCOMES:
Demographics | Baseline
  Age, gender, level of education, ethnicity, nature and frequency of any MHFA interventions directly experienced)
Change in Employees Help Seeking Intentions | Baseline, 6, 12 and 24 months.
  Employees Help seeking intentions measured by the General Help-Seeking Questionnaire [GHSQ] (Wilson et al, 2005). The GHSQ assesses future help-seeking intentions and recent and past help-seeking experiences. Intentions are measured by listing a number of potential help sources and asking employees to indicate how likely it is that they would seek help from that source for a specified problem on a 7-point scale ranging from (1) extremely unlikely to seek help to (7) extremely likely to seek help.
Change in Employees' Mental Health and Well-being | Baseline, 6, 12 and 24 months.
  Measured using the Warwick-Edinburgh Mental Health and Well-being Scale [WEMHWBS] (Tennant et al., 2007). The WEMWBS is a 14- item scale measuring mental well-being in general populations with 5 response categories: 1: none of the time to 5: all of the time in response to items such as I've been feeling optimistic about the future. Responses are summed to provide a single score ranging from 14-70. Higher scores indicate greater levels of Mental health and Wellbeing.
Change in Mental Health First-Aiders' Mental Health Literacy | Baseline, 1, 6, 12 and 24 months.
  Measured by the Mental Health Literacy Scale [MHLS], (O'Connor & Casey, 2015). The MHLS is a 35-item measure of mental health literacy - people's knowledge and beliefs of the recognition, management and prevention of mental disorders. Each item seeks a correct answer to each question with higher scores indicating higher levels of literacy.
Change in Employees' Quality of Life | Baseline, 6, 12 and 24 months.
  Measured using using the EQ-5D (Byford, 2013). The EQ-5D is a standardised measure of health-related quality of life (HRQoL) that provides a simple, generic measure of health for clinical and economic appraisal. The EQ-5D comprises five questions on mobility, self-care, pain, usual activities, and psychological status. For each question, there are 5 possible responses, ranging from best to worse. Possible scores for the EQ-5D-5 L range from 1 to - 0.594. On this scale it is considered equal to full health and 0 is equal to death. The scoring system allows for some health states to be considered 'worse than death'.
Change in Employees' Self-Efficacy for Seeking Mental Health Care | Baseline, 6, 12 and 24 months.
  Measured using the Employees' Self-Efficacy for Seeking Mental Health Care Scale [SE-SMHC] (Moore et al, 2015 adapted by Umubeyi et al, 2016).The SE-SMHC is a nine-item measure of recipients' confidence in seeking mental health care and comprises two sub-scales scales: one measuring confidence in knowing how to access mental health care and how to communicate with health care staff (SE-Knowledge), and successfully coping with the social and interpersonal consequences of seeking care (SE-Coping). The SE-SMHC is scored by asking employees to rank items from 1-10 and summed to determine low (1-3), medium (4-6) or high (7-10) confidence.
Change in Employees Social well-being | Baseline, 6, 12 and 24 months.
  Measured using the Social Well-being Scale [SWBS] (Keyes, 1998). The SWBS is a 15-item scale measuring five dimensions of social well-being, namely Social Coherence, Social Integration, Social Contribution, Social Actualisation and Social Acceptance. Participants respond to items such as "People do not care about other people's problems using a seven-point scale from strongly agree to strongly disagree which are summed for each dimension with a higher score representing greater social wellbeing.
Change in Employees' use of standard mental health and other services | Baseline, 6, 12 and 24 months.
  An adapted version of the Client Services Receipt Inventory [CSRI] (Beecham & Knapp, 2001). The CSRI gathers information on service utilisation, income, accommodation and other cost-related variables. It also captures resource use patterns and support costs to be estimated using an appropriate unit cost.
Change in Employees' Quality of Life | Baseline, 6, 12 and 24 months.
  Measured using the Short Form-12 Health Survey, [SF-12] (Ware et al, 1996). The SF-12 is 12 item standardised measure that assesses limitations in role functioning as a result of physical and mental health. A shorter form of the SF-36, the SF-12 has been used with a variety of clinical and non-clinical populations and captures eight domains of physical and mental health. Each item is scored from 1 (all of the time) to 5 (none of the time) in response to statements such as In the past four weeks, how much of the time has your physical or emotional problems interfered with your social activities? The key scores for the SF-12 are a physical health composite score (PCS-12) and a mental health score (MCS-12). Higher scores indicate higher levels of health.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Callaghan, PhD, Principal Investigator — London South Bank University
Locations (1):
- London South Bank University, London, United Kingdom

REFERENCES:
- [Derived] Atanda O, Callaghan P, Carter T, Durcan G, O'Shea N, Brown SD, Reavey P, Vangeli E, White S, Wood KV. Evaluation of Mental Health First Aid from the Perspective Of Workplace End UseRs-EMPOWER: protocol of cluster randomised trial phase. Trials. 2020 Aug 14;21(1):715. doi: 10.1186/s13063-020-04636-0. PMID 32795364